CLINICAL TRIAL: NCT04737551
Title: Adjuvant Chemoradiation Following Radical Resection of Pancreatic Ductal Adenocarcinoma, a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-RPC
Record Dates: First submitted 2021-01-25; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Resectable Pancreatic Cancer; Adjuvant Chemoradiotherapy; Surgery
MeSH Terms: interventions — Chemotherapy, Adjuvant; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No adjuvant treatment: Pancreatic cancer patients who received surgery without subsequent adjuvant treatment.
  Interventions: Other: Follow-up only
- Adjuvant chemotherapy: Pancreatic cancer patients who received surgery and only adjuvant chemotherapy.
  Interventions: Drug: Adjuvant chemotherapy
- Adjuvant chemoradiotherapy: Pancreatic cancer patients who received surgery and only adjuvant chemoradiotherapy.
  Interventions: Radiation: Adjuvant chemoradiotherapy
- Adjuvant chemoradiotherapy + adjuvant chemotherapy: Pancreatic cancer patients who received surgery and both adjuvant chemoradiotherapy and chemotherapy.
  Interventions: Radiation: Adjuvant chemoradiotherapy + Adjuvant chemotherapy

INTERVENTIONS:
Other: Follow-up only — Only routine follow-up but no treatment
  Groups: No adjuvant treatment
Drug: Adjuvant chemotherapy — Chemotherapy regimens will be decided by physicians or MDT teams, basing on patients' physical status, income status, and/or desire. Toxicity was evaluated every cycle and efficacy was evaluated every two cycles. The treatment course of adjuvant chemotherapy was followed the recommendation of NCCN guideline.
  Groups: Adjuvant chemotherapy
Radiation: Adjuvant chemoradiotherapy — Adjuvant CRT could be delivered before or simultaneously with adjuvant chemotherapy. Radiation used 6 MV or 15 MVX-ray beams delivering daily fractions of 180-200cGy to a total dose of 45-55Gy in 25-28 fractions using CT-based, three-dimensional conformal radiation therapy (3DRT), intensity-modulated radiation therapy (IMRT) or tomotherapy (TOMO).
  S-1 was administered orally at a dose of 40mg twice a day during radiation day as radiosensitizer through radiotherapy. Antiemetic medications and proton pump inhibitor were prophylactic used to reduce the occurrence of nausea and inhibit gastric acid secretion.
  Groups: Adjuvant chemoradiotherapy
Radiation: Adjuvant chemoradiotherapy + Adjuvant chemotherapy — See as above (adjuvant chemotherapy and adjuvant chemoradiotherapy).
  Groups: Adjuvant chemoradiotherapy + adjuvant chemotherapy

SUMMARY:
This is a prospective observation cohort study to evaluate efficacy of different types of adjuvant therapy strategies, including chemoradiotherapy, chemotherapy alone, or no adjuvant treatment, for pancreatic ductal adenocarcinoma patients who received surgical resection of primary cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 90 years.
2. Received surgical resection of primary tumor.
3. Histological diagnosis of pancreatic ductal adenocarcinoma.
4. Signed informed consent.

Exclusion Criteria:

1.Active concomitant malignancy (Malignancy other than pancreatic cancer).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elegible patients were those who received surgical resection of primary pancreatic tumor and were histologically diagonsed as pancreatic ductal adenocarcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to 60 months
  Overall survival (OS) was defined as the time interval from the date of surgery to the date of death due to any cause or the date a patient was last known to be alive. Estimated by using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Disease Free Survival | Up to 48 months
  Disease free survival (DFS) was defined as the time interval from the date of surgery to the date of disease recurrence or death or the date of a participant was last known to be alive without disease recurrence. Response was evaluated according to revised Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
Number of Participants Experiencing Adverse Events | Up to 60 months
  Number of participants experiencing adverse events during chemoradiation and during adjuvant chemotherapy, at any grade, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0. This is used to determine the Toxicity profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Uesaka K, Boku N, Fukutomi A, Okamura Y, Konishi M, Matsumoto I, Kaneoka Y, Shimizu Y, Nakamori S, Sakamoto H, Morinaga S, Kainuma O, Imai K, Sata N, Hishinuma S, Ojima H, Yamaguchi R, Hirano S, Sudo T, Ohashi Y; JASPAC 01 Study Group. Adjuvant chemotherapy of S-1 versus gemcitabine for resected pancreatic cancer: a phase 3, open-label, randomised, non-inferiority trial (JASPAC 01). Lancet. 2016 Jul 16;388(10041):248-57. doi: 10.1016/S0140-6736(16)30583-9. Epub 2016 Jun 2. PMID 27265347
- [Background] Goodman KA, Regine WF, Dawson LA, Ben-Josef E, Haustermans K, Bosch WR, Turian J, Abrams RA. Radiation Therapy Oncology Group consensus panel guidelines for the delineation of the clinical target volume in the postoperative treatment of pancreatic head cancer. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):901-8. doi: 10.1016/j.ijrobp.2012.01.022. Epub 2012 Apr 5. PMID 22483737
- [Background] Palta M, Godfrey D, Goodman KA, Hoffe S, Dawson LA, Dessert D, Hall WA, Herman JM, Khorana AA, Merchant N, Parekh A, Patton C, Pepek JM, Salama JK, Tuli R, Koong AC. Radiation Therapy for Pancreatic Cancer: Executive Summary of an ASTRO Clinical Practice Guideline. Pract Radiat Oncol. 2019 Sep-Oct;9(5):322-332. doi: 10.1016/j.prro.2019.06.016. PMID 31474330
- [Background] Ma SJ, Hermann GM, Prezzano KM, Serra LM, Iovoli AJ, Singh AK. Adjuvant chemotherapy followed by concurrent chemoradiation is associated with improved survival for resected stage I-II pancreatic cancer. Cancer Med. 2019 Mar;8(3):939-952. doi: 10.1002/cam4.1967. Epub 2019 Jan 16. PMID 30652417
- [Background] Abrams MJ, Huber KE, Knisely JP, Chang BW, Russo SM, Saif MW. Capecitabine as a Radiosensitizer in Adjuvant Chemoradiotherapy for Pancreatic Cancer: A Retrospective Study. Anticancer Res. 2015 Dec;35(12):6901-7. PMID 26637914